CLINICAL TRIAL: NCT04302428
Title: Zinc Status and Growth in Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Sarah Bauer, Assistant Professor, School of Medicine, Indiana University
Other Study IDs: 1907847033
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Cystic; Fibrosis
Keywords: Zinc; Growth; Nutrition; Cystic; Fibrosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric CF Patients: Pediatric patients ages 3 months to 3 years with CF identified via newborn screening.
  Interventions: Biological: Serum Zn; Biological: Red Blood Cell Zn

INTERVENTIONS:
Biological: Serum Zn — The investigators will obtain an additional 2 mL of blood in an extra tube. This will be collected at the same time blood is collected for the participant's yearly CF screening labs so as to minimize additional needle sticks.
Biological: Red Blood Cell Zn — If the participant is greater or equal than 5 kg, an additional 2 mL of blood will be obtained in an extra tube. This will be collected at the same time blood is collected for the participant's yearly CF screening labs so as to minimize additional needle sticks.

SUMMARY:
The purpose of this study is to improve the understanding of the relationship of zinc status and growth in infants and young children who were diagnosed with cystic fibrosis via newborn screening.

DETAILED DESCRIPTION:
The objective of this study is to improve the understanding of the relationship of zinc (Zn) status and growth in infant and young people with cystic fibrosis (PWCF). The investigators hypothesize that Zn deficiency in infant and young PWCF is associated with poor growth.

Aim #2: To study the association between Zn levels in red blood cells and nutritional status in PWCF at 3 months to 3 years of age and compare it to the association between serum Zn and nutritional status in the same population. Hypothesis: Lower Zn levels in red blood cells is associated with poorer nutritional status in infant and young PWCF and is a better measure of Zn status compared to serum Zn.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients ages 3 months to 3 years with CF identified via new born screening

Exclusion Criteria:

* History of meconium ileus
* History of prematurity (born prior to completing 36 weeks 6 days gestation)

Ages: 3 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients ages 3 months to 3 years with CF identified via new born screening
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Zinc Status | 1 day
  Zn status in infant and young PWCF as measured by serum Zn and red blood cell Zn

CONTACTS AND LOCATIONS:
Overall Officials: Clement Ren, MD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No